CLINICAL TRIAL: NCT00002707
Title: A RANDOMIZED TRIAL COMPARING PREOPERATIVE DOXORUBICIN (ADRIAMYCIN)/CYCLOPHOSPHAMIDE (AC) TO PREOPERATIVE AC FOLLOWED BY PREOPERATIVE DOCETAXEL (TAXOTERE) AND TO PREOPERATIVE AC FOLLOWED BY POSTOPERATIVE DOCETAXEL IN PATIENTS WITH OPERABLE CARCINOMA OF THE BREAST
Brief Title: Chemotherapy in Treating Women With Breast Cancer That Can Be Surgically Removed
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NSABP Foundation Inc (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Norman Wolmark, MD, NSABP Foundation, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NSABP B-27; CDR0000064521
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2010-02-03 (Estimated); Status verified 2010-02

CONDITIONS: Breast Cancer
Keywords: stage I breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel; Doxorubicin; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 2 (Experimental): doxorubicin and cyclophosphamide plus Taxotere prior to surgery plus tamoxifen
  Interventions: Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Doxorubicin; Drug: Tamoxifen
- Group 3 (Experimental): doxorubicin and cyclophosphamide followed by surgery followed by taxotere plus tamoxifen
  Interventions: Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Doxorubicin; Drug: Tamoxifen
- Group 1 (Active Comparator): doxorubicin and cyclophosphamide plus tamoxifen
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Tamoxifen

INTERVENTIONS:
Drug: Cyclophosphamide — 600 mg/m2 IV every 21 days for 4 cycles
Drug: Docetaxel — 100 mg/m2 IV every 21 days for 4 cycles
  Arms: Group 2; Group 3
Drug: Doxorubicin — 60 mg/m2 IV every 21 days fo 4 cycles
Drug: Tamoxifen — 20 mg p.o. once daily for 5 years starting on day 1 of ther first AC cycle

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known if chemotherapy given before surgery is more effective with or without docetaxel given before or after surgery for breast cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of chemotherapy using doxorubicin and cyclophosphamide with or without docetaxel in treating women who have stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare overall and disease-free survival in patients with operable adenocarcinoma of the breast treated with 4 courses of preoperative doxorubicin and cyclophosphamide (AC) alone vs 4 courses of preoperative or postoperative docetaxel (TXT) following 4 courses of preoperative AC. II. Evaluate whether the addition of preoperative TXT to preoperative AC results in improved rates of clinical and pathologic locoregional tumor response. III. Assess whether the addition of preoperative TXT to preoperative AC results in improved rates of breast conservation. IV. Assess whether postoperative TXT improves disease-free and overall survival in patients who receive preoperative AC, especially in certain subgroups of patients (e.g., those with pathologically positive nodes).

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to age (under 50 vs 50 and over), clinical tumor size (less than 2.1 cm vs 2.1-4.0 cm vs greater than 4.0 cm), clinical nodal status (negative vs positive), and participating center. Patients are randomized to one of three treatment arms. Arm I: Patients receive doxorubicin IV followed by cyclophosphamide IV over 30 minutes to 2 hours on day 1 every 21 days for 4 courses. Patients receive oral tamoxifen daily for 5 years, starting on day 1. After completion of chemotherapy, patients are offered surgery (e.g., lumpectomy with axillary node dissection, or modified radical mastectomy). Post-operative radiotherapy is given post-lumpectomy. Arm II: Patients receive doxorubicin IV followed by cyclophosphamide IV over 30 minutes to 2 hours followed by docetaxel IV over 1 hour on day 1 once every 21 days for 4 courses. Patients receive oral tamoxifen daily for 5 years, starting on day 1. After the completion of chemotherapy, surgery is offered (as in arm I). Radiotherapy follows surgery in post-lumpectomy patients. Arm III: Patients receive doxorubicin IV followed by cyclophosphamide IV over 30 minutes to 2 hours on day 1 every 21 days for 4 courses. Patients receive oral tamoxifen daily for 5 years, starting on day 1. After completion of chemotherapy, surgery is offered (as in arm I). After surgical recovery, docetaxel IV is given over 1 hour once every 21 days for 4 courses. Radiotherapy follows docetaxel in post-lumpectomy patients. Chemotherapy is repeated every 21 days for 4 courses in the absence of disease progression or unacceptable toxicity. Patients are followed every 6 months for 5 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 2,400 patients will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically proven invasive adenocarcinoma of the breast Fine-needle aspiration is acceptable Core or Tru-cut biopsies are preferable No more than 63 days between initial diagnosis and randomization Tumor palpable on clinical exam and confined to the breast and ipsilateral axilla If clinically negative axillary nodes (N0): primary tumor greater than 1 cm (T1c-T3) If clinically positive axillary nodes (N1): any size primary tumor (T1-3) No N2 disease, i.e., ipsilateral nodes clinically fixed to one another or to other structures No skeletal pain unless: Bone scan and/or roentgenologic exam negative for metastatic disease Suspicious findings confirmed as benign by x-ray, MRI, or biopsy No ulceration, erythema, skin infiltration (complete fixation), or peau d'orange, or skin edema of any magnitude Tethering or dimpling of skin or nipple inversion allowed No bilateral malignancy Suspicious contralateral mass proven benign on biopsy allowed None of the following unless proven benign on biopsy: Suspicious palpable nodes in contralateral axilla Palpable supraclavicular or infraclavicular nodes Hormone receptor status: Any status

PATIENT CHARACTERISTICS: Age: Any age Sex: Female Menopausal status: Not specified Performance status: Not specified Life expectancy: At least 10 years (exclusive of cancer diagnosis) Hematopoietic: WBC at least 4,000/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin normal AST/ALT normal Alkaline phosphatase normal Renal: Creatinine normal Cardiovascular: No active cardiac disease that would preclude doxorubicin, e.g.: Documented myocardial infarction History of congestive heart failure Angina pectoris requiring medication Valvular disease with documented cardiac function compromise Arrhythmia associated with heart failure or cardiac dysfunction Poorly controlled hypertension, i.e., diastolic blood pressure greater than 100 mm Hg Cardiomegaly on chest x-ray or ventricular hypertrophy on EKG unless left ventricular ejection fraction at least 45% by MUGA Other: No other malignancy within the past 10 years except: Segmentally resected lobular carcinoma in situ of the ipsilateral or contralateral breast Effectively treated nonmelanomatous skin cancer Surgically treated carcinoma in situ of the cervix No systemic disease that would preclude therapy No psychiatric or addictive disorder that would preclude informed consent Geographically accessible for follow-up Not pregnant

PRIOR CONCURRENT THERAPY: No prior therapy for breast cancer No prior anthracyclines for any malignancy No concurrent sex hormones (e.g., birth control pills or ovarian replacement therapy)

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2411 (Actual)
Dates: Start 1995-12; Primary Completion 2002-06 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Determine if 4 cycle of pre-op or post-op Taxotere given after 4 cycles of pre-op AC will more effectively prolong survival (S) than does 4 cycles of pre-op AC alone. | Time from randomization to death from any cause.

SECONDARY OUTCOMES:
Prolonging disease-free survival (DFS). | Time from randomization to first related event of inoperable disease; residual disease following surgery; local, regional or distant recurrence; second primary cancer; death from any cause other than cancer.
Clinical loco-regional tumor response to preoperative chemotherapy. | 3-4 weeks after the last cycle of pre-op chemotherapy.
Pathologic loco-regional tumor response to pre-op chemotherapy. | At time of surgery.
Breast conservation assessment. | Assessed following surgery.
Evaluate if post-op Taxotere is of benefit in patients who received pre-op AC and, if so, whether it is of benefit in certain subgroups of patients. | DFS and S will be assessed in patient subgroups.

CONTACTS AND LOCATIONS:
Overall Officials: Harry D. Bear, MD, PhD, Study Chair — Massey Cancer Center
Locations (145):
- United States (134):
  - Huntsville Hospital System, Huntsville, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Sutter Health Western Division Cancer Research Group, Greenbrae, California
  - Loma Linda University Medical Center, Loma Linda, California
  - Saint Mary Medical Center - Long Beach, Long Beach, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Comprehensive Cancer Centers of the Desert, Palm Springs, California
  - Kaiser Permanente-Southern California Permanente Medical Group, San Diego, California
  - Catholic Healthcare West - Westbay Region, San Francisco, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - CCOP - Colorado Cancer Research Program, Inc., Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - CCOP - Christiana Care Health Services, Wilmington, Delaware
  - George Washington University Cancer Center, Washington D.C., District of Columbia
  - Halifax Medical Center, Daytona Beach, Florida
  - Baptist Regional Cancer Institute - Jacksonville, Jacksonville, Florida
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - CCOP - Mount Sinai Medical Center, Miami Beach, Florida
  - Good Samaritan Medical Center, West Palm Beach, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Medical College of Georgia Comprehensive Cancer Center, Augusta, Georgia
  - Dwight David Eisenhower Army Medical Center, Fort Gordon, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - North Idaho Cancer Center, Coeur d'Alene, Idaho
  - Illinois Masonic Medical Center, Chicago, Illinois
  - CCOP - Evanston, Evanston, Illinois
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - Rockford Clinic, Rockford, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - St. Vincent Hospital and Health Care Center, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Lucille Parker Markey Cancer Center, University of Kentucky, Lexington, Kentucky
  - Norton Healthcare System, Louisville, Kentucky
  - Louisiana State University Medical Center - New Orleans, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - CCOP - Ochsner, New Orleans, Louisiana
  - Eastern Maine Medical Center, Bangor, Maine
  - Franklin Square Hospital Center, Baltimore, Maryland
  - National Naval Medical Center, Bethesda, Maryland
  - Regional Cancer Therapy Center - Frederick, Frederick, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Lahey Clinic - Burlington, Burlington, Massachusetts
  - Berkshire Medical Center, Pittsfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Michigan State University, East Lansing, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Ellis Fischel Cancer Center - Columbia, Columbia, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University School of Medicine, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Methodist Cancer Center - Omaha, Omaha, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - CCOP - Southern Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Cooper Cancer Institute, Camden, New Jersey
  - Trinitas Hospital - Jersey Street Campus, Elizabeth, New Jersey
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - University of Medicine and Dentistry of New Jersey, Newark, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico
  - CCOP - Syracuse Hematology-Oncology Associates of Central New York, P.C., Syracuse, New York
  - Lineberger Comprehensive Cancer Center, UNC, Chapel Hill, North Carolina
  - East Carolina University School of Medicine, Greenville, North Carolina
  - CCOP - Southeast Cancer Control Consortium, Winston-Salem, North Carolina
  - Comprehensive Cancer Center of Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Akron City Hospital, Akron, Ohio
  - Aultman Cancer Center, Canton, Ohio
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Jewish Hospital of Cincinnati, Inc., Cincinnati, Ohio
  - South Pointe Hospital, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - CCOP - Sooner State, Tulsa, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - St. Luke's Network - Bethlehem, Bethlehem, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Kent County Memorial Hospital - Rhode Island, Warwick, Rhode Island
  - Medical University of South Carolina, Charleston, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - CCOP - Baptist Cancer Institute, Memphis, Tennessee
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Medical Group of Texas, Dallas, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Baylor College of Medicine, Houston, Texas
  - Joe Arrington Cancer Research and Treatment Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - CCOP - Southwestern Vermont Regional Cancer Center, Bennington, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Virginia Oncology Associates, Newport News, Virginia
  - Eastern Virginia Medical School, Norfolk, Virginia
  - MBCCOP - Massey Cancer Center, Richmond, Virginia
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington
  - David Lee Cancer Center, Charleston, West Virginia
  - West Virginia University Hospitals, Morgantown, West Virginia
  - Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - St. Vincent Hospital, Green Bay, Wisconsin
  - CCOP - Marshfield Medical Research and Education Foundation, Marshfield, Wisconsin
  - St. Luke's Medical Center, Milwaukee, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (11):
  - Tom Baker Cancer Center - Calgary, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Credit Valley Hospital, Mississauga, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - Royal Victoria Hospital - Montreal, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec
  - Jewish General Hospital - Montreal, Montreal, Quebec
  - St. Mary's Hospital Center, Montreal, Quebec
  - Hopital du Saint-Sacrament, Quebec, Québec, Quebec
  - L'Hopital Laval, Ste-Foy, Quebec

REFERENCES:
- [Background] Rastogi P, Anderson SJ, Bear HD, Geyer CE, Kahlenberg MS, Robidoux A, Margolese RG, Hoehn JL, Vogel VG, Dakhil SR, Tamkus D, King KM, Pajon ER, Wright MJ, Robert J, Paik S, Mamounas EP, Wolmark N. Preoperative chemotherapy: updates of National Surgical Adjuvant Breast and Bowel Project Protocols B-18 and B-27. J Clin Oncol. 2008 Feb 10;26(5):778-85. doi: 10.1200/JCO.2007.15.0235. PMID 18258986
- [Background] Soran A, Nesbitt L, Mamounas EP, Lembersky B, Bryant J, Anderson S, Brown A, Passarello M. Centralized medical monitoring in phase III clinical trials: the National Surgical Adjuvant Breast and Bowel Project (NSABP) experience. Clin Trials. 2006;3(5):478-85. doi: 10.1177/1740774506070747. PMID 17060221
- [Background] Heys SD, Sarkar T, Hutcheon AW. Primary docetaxel chemotherapy in patients with breast cancer: impact on response and survival. Breast Cancer Res Treat. 2005 Mar;90(2):169-85. doi: 10.1007/s10549-004-1001-0. PMID 15803364
- [Result] Bear HD, Anderson S, Smith RE, Geyer CE Jr, Mamounas EP, Fisher B, Brown AM, Robidoux A, Margolese R, Kahlenberg MS, Paik S, Soran A, Wickerham DL, Wolmark N. Sequential preoperative or postoperative docetaxel added to preoperative doxorubicin plus cyclophosphamide for operable breast cancer:National Surgical Adjuvant Breast and Bowel Project Protocol B-27. J Clin Oncol. 2006 May 1;24(13):2019-27. doi: 10.1200/JCO.2005.04.1665. Epub 2006 Apr 10. PMID 16606972
- [Result] Julian T, Anderson S, Fourchotte V, et al.: Is invasive lobular breast cancer a prognostic factor for neoadjuvant chemotherapy response and long term outcomes? [Abstract] Breast Cancer Res Treat 100 (Suppl 1): A-3065, S146, 2006.
- [Result] Mamounas EP, Brown A, Anderson S, Smith R, Julian T, Miller B, Bear HD, Caldwell CB, Walker AP, Mikkelson WM, Stauffer JS, Robidoux A, Theoret H, Soran A, Fisher B, Wickerham DL, Wolmark N. Sentinel node biopsy after neoadjuvant chemotherapy in breast cancer: results from National Surgical Adjuvant Breast and Bowel Project Protocol B-27. J Clin Oncol. 2005 Apr 20;23(12):2694-702. doi: 10.1200/JCO.2005.05.188. PMID 15837984
- [Result] Bear HD, Anderson S, Smith RE, et al.: A randomized trial comparing preoperative (preop) doxorubicin/cyclophosphamide (AC) to preop AC followed by preop docetaxel (T) and to preop AC followed by postoperative (postop) T in patients (pts) with operable carcinoma of the breast: results of NSABP B-27. [Abstract] Breast Cancer Res Treat 88 (Suppl 1): A-26, 2004.
- [Result] Bear HD, Anderson S, Brown A, Smith R, Mamounas EP, Fisher B, Margolese R, Theoret H, Soran A, Wickerham DL, Wolmark N; National Surgical Adjuvant Breast and Bowel Project Protocol B-27. The effect on tumor response of adding sequential preoperative docetaxel to preoperative doxorubicin and cyclophosphamide: preliminary results from National Surgical Adjuvant Breast and Bowel Project Protocol B-27. J Clin Oncol. 2003 Nov 15;21(22):4165-74. doi: 10.1200/JCO.2003.12.005. Epub 2003 Oct 14. PMID 14559892
- [Result] Mamounas EP, Brown A, Smith R, et al.: Accuracy of sentinel node biopsy after neoadjuvant chemotherapy in breast cancer: updated results from NSABP B-27. [Abstract] Proceedings of the American Society of Clinical Oncology 21: A-140, 2002.